CLINICAL TRIAL: NCT02137954
Title: Efficacy of Lidocaine Versus Placebo in Palliative Care Patients With Opioid-refractory Cancer Pain With Neuropathic Component: a Multicenter, Prospective, Double-blind Randomized Placebo-controlled Study.
Acronym: LIDOSP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-50
Record Dates: First submitted 2014-05-07; First posted 2014-05-14 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Cancer; Pain With Neuropathic Component
Keywords: cancer; pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine (Active Comparator): Lidocaine. Initial dose IV will be 5 mg/kg per day during the first 24 hours the 8 mg/kg per day
  Interventions: Drug: Lidocaine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine
  Other Names: Lidocaine. Initial dose IV will be 5 mg/kg per day during the first 24 hours the 8 mg/kg per day
  Arms: lidocaine
Drug: Placebo
  Arms: placebo

SUMMARY:
This is a multicenter, prospective, randomized, placebo-controlled, double-blind, two-parallel groups study comparing lidocaine (experimental group) to placebo (control group). The study protocol was elaborated using the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) Statement.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient suffering from cancer pain refractory to standard opiates (numeric pain intensity scale NPIS >=4/10 after 24 hours of continuous intravenous morphine or oxycodone administration [SOR 2002, analgesics drugs for adults cancer nociceptive pain]), regardless of the nature of the primary cancer]
* Patient suffering from cancer neuropathic or mixed pain (DNA survey score> = 4 [Bouhassira 2004])
* Patient receiving palliative care as defined by French Society of Palliative and Support Care [Charte des Soins Palliatifs, 1996, Act No. 99-477 of 9 June 1999 to guarantee the right of access to palliative care] according to the definition of the World Health Organization (WHO) [World Health Organization. WHO's pain ladder. http://www.who.int/cancer/palliative/painladder/en/. Accessed December 9.2011]
* Patient with histological diagnosis of cancer, locally advanced or metastatic disease
* Patient without curative cancer treatment, and with or without palliative anticancer treatment
* Patient hospitalized in a specific palliative care unit
* Patient with an estimated survival higher than 48 hours (physician estimation) Patient providing written informed consent for participation prior to any study procedures.

Exclusion Criteria:

* Patient with a known hypersensitivity to lidocaine
* Patient with a history of porphyria, arrhythmias, disorders of atrioventricular conduction requiring permanent pacing not yet realized, uncontrolled epilepsy, uncontrolled hypertension
* Patient with hematologic malignancy, abnormal renal, hepatic and cardiac functions
* Patient with a altered sleepiness (Epworth scale score ≤ 16)
* Patient with altered cognitive function (TELECOM scale score> 11) [Arsène 2000]
* Patient not native French speaker Patient defined as vulnerable subject (minor subject, pregnant or nursing woman, subject freedom deprived)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficacy | 40 minutes
  Analgesic efficacy will be assessed from several endpoints. The primary endpoint will be defined as the change of pain level between baseline (T0) and 40 minutes (T1) after baseline. The pain level will be assessed using a self-administered numeric pain intensity scale (NPIS), ranged from 0 (no pain) to 10 (worst pain possible). A minimal 30% decrease of pain level between baseline and T1 will define the success, and other cases will define the failure of the treatment.

SECONDARY OUTCOMES:
intensity of the pain neuropathic | 120 minutes
  the intensity of the pain neuropathic component using the Neuropathic Pain Symptom Inventory (NPSI) at T4, T5, and T6 {Bouhassira, 2004 #9}; the NPSI is a 12-item self-administered questionnaire describing the intensity of the symptoms associated with pain neuropathic

OTHER OUTCOMES:
raw values of pain levels (NPIS) | 40 minutes
  raw values of pain levels (NPIS) at each evaluation time, percentage of reduction between the initial level of pain and other evaluation times
tolerance to the treatments | 48 hours
  The tolerance to the treatment (lidocaine) will be assessed during the first 48 hours following the treatment administration. Adverse events will be cautiously collected (intensity and discomfort): i) lidocaine: arrhythmia, blurred vision, headache, malaise, tremors, metallic taste, nausea/vomiting, perioral numbness and tingling, sedation, and tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien SALAS, MD, Principal Investigator — - Service d'Oncologie Médicale et de Soins Palliatifs Assistance Publique Hopitaux de Marseille
Locations (1):
- - Service d'Oncologie Médicale et de Soins Palliatifs Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Salas S, Auquier P, Duffaud F, Garnier SR, Deschamps M, Honore S, Sudour P, Baumstarck K. Efficacy of lidocaine in patients receiving palliative care with opioid-refractory cancer pain with a neuropathic component: study protocol for a randomized controlled study. Trials. 2014 Aug 12;15:318. doi: 10.1186/1745-6215-15-318. PMID 25112302